CLINICAL TRIAL: NCT02541227
Title: Cerebrolysin REGistry Study in Stroke A Registry Study to Assess Practices, Safety and Effectiveness of Cerebrolysin in Routine Treatment of Acute Ischemic Stroke
Brief Title: Cerebrolysin REGistry Study in Stroke
Acronym: CREGS-S
Status: Terminated | Type: Observational
Why Stopped: The goal to match 1000 patients per group could not be achieved with reasonable effort and in reasonable time.
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: SITS International (Network)
Responsible Party: Sponsor
Other Study IDs: EVER-GB-0514
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cerebrolysin group: Patients who are treated with Cerebrolysin; dosage, frequency and duration follows local clinical practice in accordance with the terms of the local marketing authorization
  Interventions: Drug: Cerebrolysin
- Control group: Patients who are not treated with Cerebrolysin; treatment follows local clinical practice

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin dosage, frequency and duration follows local clinical practice in accordance with the terms of the local marketing authorization
  Groups: Cerebrolysin group

SUMMARY:
Investigation of clinical practices, safety and effectiveness of Cerebrolysin in routine treatment of patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Stroke is a devastating disease and one of the primary causes for death and long term morbidity imposing a heavy burden on patients, relatives and the health care system. Except for fibrinolytic therapy, which is only possible in a minor fraction of patients, there is no widely approved medication for the treatment of acute stroke.

Cerebrolysin has been approved for the treatment of stroke in over 45 countries worldwide.

Since the approval of Cerebrolysin, stroke therapy has evolved, namely, with improved overall care, stroke units, more targeted rehabilitation, and the increasing availability of fibrinolytic therapy (rtPA, Actilyse) in specialized centers throughout the world. More recently, interventional therapies with various thrombus retrievers have emerged.

In addition the Cerebrolysin treatment in stroke has evolved with different time windows, dosages and lengths of therapy being given in a pragmatic way by physicians within the specification of Product Characteristics for Cerebrolysin (SPC). The main aim of this study is to capture these variables of the Cerebrolysin treatment and its comedication in order to give guidance to further research. This research may consist of an extension of the current registry or targeted research in one or several subgroups of patients responding to Cerebrolysin treatment.

It is therefore the overall aim of this registry study to monitor the effectiveness and safety of Cerebrolysin therapy against the background of the now established and evolving stroke therapies. In the concomitant control group these therapies alone or in combination will be compared to the addition of Cerebrolysin in these patients. Of particular interest is the treatment in stroke units, with rtPA and systematic rehabilitation.

An open observational treatment design has been chosen to collect data to capture the therapies as applied in real clinical practice and to avoid the selection bias typical for controlled studies excluding the majority of patients from participation. In order to overcome the observational bias as major and inherent limitation of open trial designs, a remote and blinded assessment will be done: after three months treatment the patients' assessment of the modified Rankin Scale (mRS, a widely accepted primary outcome parameter) will be -after specific informed consent- video-taped and subsequently assessed by at least two independent and blinded assessors experienced in the remote assessment of the mRS.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Clinical diagnosis of acute ischemic stroke
* Patient's independence prior to stroke onset (pre-morbid mRS of 0 or 1)
* Reasonable expectation of successful follow-up (max. 100 days)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receive acute ishemic stroke care according to local treatment standards, not amended or influenced by the study
Sampling Method: Probability Sample
Enrollment: 1823 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 days
  Ordinal analysis of the mRS on day 90 was chosen as statistically powerful primary endpoint, as it is robust to case mix, clinically relevant and treatment-responsive.

SECONDARY OUTCOMES:
The National Institutes of Health Stroke Scale (NIHSS) | 90 days
  Ordinal NIHSS at 3 months after stroke onset
  o Home Time (number of nights among the first 90 days after stroke onset that the patient spends in his own or a relative's private home)
Montreal Cognitive Assessment (MoCA) | 90 days
  Ordinal MoCA assessment of cognitive functions at 3 months after stroke
Home Time (number of nights among the first 90 days after stroke onset that the patient spends in his own or a relative's private home) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Kennedy Lees, MD, Study Chair — University of Glasgow
Locations (1):
- AKH Linz, Linz, Austria